CLINICAL TRIAL: NCT04035603
Title: Multimodal CET for Smoking Cessation Augmented With D-cycloserine
Brief Title: Multimodal Cue Exposure Therapy for Smoking Cessation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Never received funding
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Michael Otto, Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01DA048043
Record Dates: First submitted 2019-06-19; First posted 2019-07-29 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- D-Cycloserine Augmentation (Experimental): D-cycloserine (DCS) augmentation of CET sessions
  Interventions: Drug: D-Cycloserine; Behavioral: Open Phase CBT that preceeds the randomization phase; Drug: Open phase smoking cessation pharmacotherapy that proceeds the randomization phase
- Placebo Augmentation (Placebo Comparator): Placebo (PBO) augmentation of CET sessions
  Interventions: Drug: Placebo oral tablet; Behavioral: Open Phase CBT that preceeds the randomization phase; Drug: Open phase smoking cessation pharmacotherapy that proceeds the randomization phase

INTERVENTIONS:
Drug: D-Cycloserine — 50 mg d-cycloserine given as an augmentation agent, 70 minutes prior to three CET sessions for participants who achieved smoking cessation following open treatment.
  Other Names: DCS
  Arms: D-Cycloserine Augmentation
Drug: Placebo oral tablet — matching 50 mg identical placebo given as an augmentation agent, 70 minutes prior to three CET sessions for participants who achieved smoking cessation following open treatment.
  Other Names: PBO
  Arms: Placebo Augmentation
Behavioral: Open Phase CBT that preceeds the randomization phase — Four sessions of weekly individual cognitive-behavior therapy (CBT: a form of psychotherapy that treats problems by helping people modify thoughts, behaviors, and emotions; in this case, for the goal of smoking cessation). Session topics include educational (e.g., health risks of smoking, effectiveness of different treatment approaches), motivational enhancement (e.g., identifying personally relevant benefits of quitting, and costs of continuing to smoke), and cognitive-behavioral elements (e.g., identifying smoking triggers, developing coping strategies for these triggers, planning for high risk situations, relapse prevention).
Drug: Open phase smoking cessation pharmacotherapy that proceeds the randomization phase — Initiating 2 weeks prior to quit date and continuing for 8 weeks after quit date, choice of one of three pharmacological smoking cessation aids: Nicotine Replacement Therapy (nicotine patch), Varenicline, or Bupropion.

SUMMARY:
At two sites (Boston University and the University of Texas at Austin, under the MPI direction of Drs. Otto and Smits) the investigators propose to randomly assign 240 adult smokers who have achieved short-term abstinence following open treatment with a 4 session cognitive-behavior therapy program combined with medication (nicotine patch, varenicline, or bupropion, selected openly) to (1) d-cycloserine augmentation of multimodal cue exposure therapy (CET), or (2) placebo augmentation of multimodal CET. This Stage II project is designed to: (1) evaluate the short-term and long-term efficacy of the experimental intervention, (2) further test putative mechanisms of change, (3) explore possible moderator effects of theoretically-relevant variables, and (4) use innovative, multimodal CET strategies. Putative mediators and smoking abstinence will be assessed during the intervention period and up to 6 months following the quit attempt.

DETAILED DESCRIPTION:
This study utilizes on open phase of 4-sessions of cognitive-behavior therapy for smoking cessation that is combined with open pharmacotherapy (selected by participants in collaboration with the study medical team: nicotine patch, varenicline, or bupropion). Session topics include educational (e.g., health risks of smoking, effectiveness of different treatment approaches), motivational enhancement (e.g., identifying personally relevant benefits of quitting, and costs of continuing to smoke), and cognitive-behavioral elements (e.g., identifying smoking triggers, developing coping strategies for these triggers, planning for high risk situations, relapse prevention). The study therapists will also make a supportive phone call on the day of the quit attempt, with repeated check-in calls over the quit window (i.e., weeks 4-6) as needed for individuals having difficulties reaching abstinence. Participants who fail to achieve smoking cessation during the quit period window will be referred for clinical treatment as desired in the center the study is conducted in or an alternative site.

Following successful smoking abstinence at Week 0 (Week 0 is defined by 24 hr abstinence within a two-week grace period of the target date), participants will be randomized to the study drug condition (50 mg DCS or matching placebo) combined with cue-exposure therapy (CET). CET is manualized and will have four modalities: (1) exposure to slides of smoking (pictorial), (2) exposure to emotions and imagined situations that most reliably trigger an urge to smoke (emotional/imaginal), (3) exposure to a participant's own cigarettes and pack (in vivo),70 and (4) personalized and immersive 360° VR exposure (participants select the VR scene-e.g., break time outside work, evening party, car ride that best corresponds to their highest craving situation). CET sessions are scheduled for the quit week, one week later, and again 8 weeks later. Smoking cessation assessments continue across 24 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria: (open phase)

* daily smoker for at least one year, smoking an average of at least 10 cigarettes per day, and motivated to quit smoking (>5 on a 10 point scale)
* had reactivity to in vivo smoking cues (an increase of two points or maximal score of 10 on a 10 point visual analogue craving scale [VAS]) following no smoking for a minimum of two hours
* medical clearance to participate in the protocol

Exclusion Criteria:

* use of other tobacco products
* current unstable medical illness (i.e. deemed as at high risk of significant worsening by study intervention procedures by study physician; e.g. heart disease, chronic obstructive pulmonary disease, or seizure disorders - assessed during telephone prescreen and initial assessment), seizure disorder, pregnancy, breastfeeding, or use of isoniazid or ethionamide
* lifetime history of psychotic disorders or uncontrolled bipolar disorder, by DSM-5 criteria as assessed by the MIni International Neuropsychiatric Interview
* substance use disorder other than nicotine or caffeine active in the past 6 months, or excessive concurrent alcohol use as defined by self-report of an average of >21 standardized drinks per week for males or >14 standardized drinks per week for females
* elevated suicide risk as determined by clinician interview
* current use of any psychotropic medications or pharmacotherapy or psychotherapy for smoking cessation not provided by the investigators during the quit attempt
* known hypersensitivity to DCS
* insufficient command of the English language or inability to understand study procedures and participate in the informed consent process

To progress to the randomized phase:

* participants must achieve a 24 hour abstinence period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Rates of Prolonged Abstinence (PA) | Prolonged abstinence is assessed from Quit week to Week 24 of Follow-up
  Failure to maintain PA at any assessment will be defined by 7 or more consecutive days of smoking or smoking at least 1 cigarette over the 2 consecutive weeks prior to the assessment
Rates of Point Prevalence Abstinence (PPA) | Point Prevalence Abstinence is assessed from Quit Week to 24 week Follow-up using a growth curve model
  PPA is defined as no smoking in the 7 days prior to any assessment. Self-report is verified with saliva cotinine.

SECONDARY OUTCOMES:
Cue-Induces Patient Rating of Craving for Cigarettes | Post-quit weeks 0, 1, 2, 9, and 10
  Cravings in response to visual, in vivo, imaginal, and VR smoking cues rated according to a 0 to 11 visual analogue scale; higher scores represent higher craving levels.

IPD SHARING:
Plan to Share IPD: Yes
One year after publication of the primary aims from this project the primary and fully de-identified IPD will be made available by the investigators on CD for other researchers providing documented IRB consent from their institution.
Supporting Information: Study Protocol, Analytic Code
Time Frame: One year after publication of primary aims
Access Criteria: Institutional IRB approval